CLINICAL TRIAL: NCT04471259
Title: Functional Follow-up After Endoscopic Calcaneoplasty for Haglund's Deformity
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018151
Record Dates: First submitted 2020-06-27; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Haglund's Deformity
Keywords: Haglund's Deformity; Biodex System; Isokinetic muscle testing; Endoscopy
MeSH Terms: interventions — Statistics as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients' injured side: The Biodex, AOFAS, VAS were tested on the patients' injured side
  Interventions: Other: Classification statistics
- Patients' uninjured side: The Biodex, AOFAS, VAS were tested on the patients' uninjured side
  Interventions: Other: Classification statistics

INTERVENTIONS:
Other: Classification statistics — We classified patients by gender, age, recovery time,etc

SUMMARY:
Isokinetic muscle strength test implemented by the Biodex system is a method used for evaluating muscle function that has been applied clinically in the field of sports and rehabilitation medicine. However, information on its application on Haglund's deformity remain insufficient. Therefore, the present study is designed to examine the effectiveness of the muscle strength test using the Biodex system in evaluating the recovery of athletic capacity in patients with Haglund's deformity following endoscopic surgery.

DETAILED DESCRIPTION:
Patients. A retrospective (medical records), level 3 evidence study was designed to evaluate the outcomes of patients who underwent endoscopic surgery for Haglund's deformity. The present study was approved by the Peking University Third Hospital's ethics committee. Written informed consent was obtained from all patients, parents or guardians of the patients prior to the present study. The rights of the patients were protected.

Diagnosis. Patients were designed to be diagnosed based on subjective complaints, combined with clinical and radiological examinations. Radiological measurements for this disease include the Fowler-Phillip angle, calcaneal pith angle, parallel pitch lines, Chauveaux-Liet angle and the X/Y ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic surgery for Haglund's deformity

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 42 cases of 37 patients diagnosed with Haglund disease treated by the author from 2012 to 2018 treated with endoscopic surgery (5 of whom were patients with left and right feet, 33 men, 4 women, average age 32.3 (range:15 to 62, SD=13.6) years, 2 of whom are professional athletes.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-01-22 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Biodex results on both sides before surgery | pre-surgery
  Biodex isokinetic muscle testing system was applied in this research. Isokinetic muscle strength test is a kind of muscle function evaluation and test method, which has been applied in the research and clinical work of sports medicine and rehabilitation medicine but never on Haglund's disease before. The isokinetic muscle strength test of the flexor and dorsiflexion of the ankle joint can evaluate the muscle strength and endurance to reflect the postoperative patient's capacity for action, providing reliable clinical evidence for postoperative rehabilitation of patients after endoscopic calcaneoplasties. Isokinetic strength test conducted on both the injured and uninjured sides of the patients using the Biodex system before surgery.
Biodex results on both sides at 3 months | 3 months after surgery
  Isokinetic strength test conducted on both the injured and uninjured sides of the patients using the Biodex system 3 months after surgery.
Biodex results on both sides at 6 months | 6 months after surgery
  Isokinetic strength test conducted on both the injured and uninjured sides of the patients using the Biodex system 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No